CLINICAL TRIAL: NCT02178683
Title: Tacrolimus and Mycophenolate Mofetil as Post-Grafting Immunosuppression After Conditioning With Fludarabine and Low-Dose Total Body Irradiation for Recipients of HLA-Matched or Mis-Matched Family or Unrelated Donor HCT
Brief Title: Tacrolimus and Mycophenolate Mofetil as Post-Grafting Immunosuppression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado Blood Cancer Institute (Other)
Responsible Party: Principal Investigator, Peter McSweeney, M.D., Principal Investigator, Colorado Blood Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBCI-157
Record Dates: First submitted 2014-05-16; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Graft Versus Host Disease
Keywords: TACROLIMUS; MYCOPHENOLATE MOFETIL; FLUDARABINE; HLA-MATCHED; MIS-MATCHED
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus and Mycophenolate Mofetil (No Intervention): Non-myeloablative allogeneic SCT from an HLA-Identical or non-identical family onor or unrelated donors, with fludarabine and low-dose TBI, with immunosuppression utilizing tacrolimus and MMF.
  Interventions: Drug: Tacrolimus and MMF.

INTERVENTIONS:
Drug: Tacrolimus and MMF. — First dose of Tacrolimus is given day -4, this continues through day +365. First dose of MMF is given within 4 hours of stem cell infusion, this continues through day +365.
  Other Names: Cellcept; MYCOPHENOLATE MOFETIL

SUMMARY:
This protocol will evaluate Tacrolimus and MMF after conditioning with fludarabine and low-dose TBI in patients who are not candidates for conventional allografting. A novel approach to immunosuppression will be tested incorporating an early but extended taper of Tacrolimus starting on day +80 or in the case of relapse. The goal is to induce early immunity and GVT effects without compromising GVHD control. The anti-metabolite MMF will be re-introduced on day +100 to try and induce tolerance and block chronic GVHD during the taper of the Tacrolimus. DLI may be given in the presence of disease progression but not for mixed chimerism as in previous protocols.

DETAILED DESCRIPTION:
OBJECTIVES

Major Objectives A. To determine whether stable allogeneic hematopoietic engraftment can be safely established in patients receiving a non-myeloablative allogeneic SCT from an HLA-Identical or non-identical family donor or unrelated donors, with fludarabine and low-dose TBI, with immunosuppression utilizing tacrolimus and MMF.

B. To evaluate the incidence of grade II-IV GVHD associated with this treatment.

C. To evaluate the engraftment when donors who are not HLA-identical family members are utilized for allogeneic stem cell transplantation.

D. To evaluate the incidence of GVHD using three times per day MMF after unrelated donor stem cell transplants or two times per day MMF after family donor stem cell transplant.

Minor Objectives A. To evaluate the incidence of chronic GVHD utilizing Tac/MMF with peripheral blood stem cells from matched or mis-matched allogeneic donors.

B. To evaluate disease responses and survival after Flu/TBI allogeneic SCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML, ALL, CML, CLL, myelodysplastic syndrome (MDS), NHL, Hodgkin's disease (HD), paroxysmal nocturnal hemoglobinuria (PNH), hypoproliferative dysplasia with or without increased blasts, or myeloma, who are at significantly higher than usual risk for mortality from conventional myeloablative allogeneic SCT due to age or comorbidities:
* Age ≥ to 50 years with AML or ALL in complete remission or with <18% blasts in bone marrow
* Age ≥ to 50 years with MDS or CML.
* Age 16 to 75 years with lymphomas or myeloma, who have failed chemotherapy and are not candidates for an autologous transplant, or who have failed a prior autologous SCT.
* Patients of any age with CLL or low-grade NHL. Patients with CLL and low-grade NHL need to have failed at least first-line treatment, with an alkylating agent, fludarabine or 2-chlorodeoxyadenosine (2-CDA), or anti-CD20 monoclonal antibody rituximab.
* Patients of any age with marrow failure
* Patients ≥60 years old will first be considered for an allogeneic stem cell transplant from a family member and will be offered an unrelated donor transplant only if no suitable family member, preferably an HLA-matched sibling, is available.
* Patients with hematological malignancy relapsed after prior auto transplantation.
* Patients at high-risk (>60%) of relapsing after autologous transplantation for hematological malignancies may receive allogeneic transplant as "consolidative immunotherapy". Diagnoses include MM, non-HL, HL, AML, ALL and MDS. Minimal duration between auto and allo transplants is 4 weeks.
* Patients of any age with hematologic malignancies treatable by allo SCT, who, because of pre-existing medical conditions or the disease itself (Fanconi anemia or PNH), are considered to be at significantly increased risk for transplant toxicity using high-dose transplantation regimens.
* Patients with metastatic renal cell carcinoma. Must have include good performance status (Karnofsky score ≥ 60%), no active brain metastases, life expectancy of at least 6 months, absence of bulky liver metastases. Patients will be treated on other active disease-specific protocols when available.
* Patients with other malignant diseases treatable with allogeneic SCT may be eligible for this protocol on a case by case basis, if approved by the principal investigator and the BMT attending physicians group.
* Available HLA-identical, a one-antigen mis-matched sibling donor, a phenotypically HLA-matched family member, a phenotypically matched unrelated donor, or a 9/10 matched unrelated donor.
* Age ≤ 75 years.

Exclusion Criteria:

* Patients with hematological malignancies eligible for a curative autologous SCT: intermediate- or high-grade NHL with chemo-sensitive first relapse.
* HD with chemo-sensitive first relapse.
* Otherwise healthy patients who are eligible for a conventional myeloablative allogeneic SCT.
* Patients with rapidly progressive intermediate or high-grade NHL, unless in minimal disease state after the last treatment.
* Patients with active uncontrolled CNS involvement with malignancy.
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment.
* Females who are pregnant.
* Patients who are HIV positive
* Organ dysfunction

  * Left ventricle ejection fraction < 35%.
  * DLCO <35% of predicted, or receiving continuous supplementary oxygen.
  * Liver function tests: total bilirubin >2x the upper limit of normal, and/or transaminases >4x the upper limit of normal.
  * Karnofsky score <50 for patients < 60 years, or <70 for patients aged 60 - 69 years
  * Creatinine clearance < 60 ml/min.
  * Patients with hypertension that is poorly controlled on antihypertensive therapy.
  * Patients with a positive PRA or anti-donor T or B cell (+) will be considered for this treatment protocol only if no other option is available.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Engraftment | Post 100 days
  To measure safe, stable engraftment using Tacrolimus and Mycophenolate Mofetil as post-grafting immunosuppression in patients following conditioning with fludarabine and total-body irradiation for allogeneic stem cell transplant.

SECONDARY OUTCOMES:
Graft Versus Host Disease | Post 100 days
  To measure the incidence of grade II-IV GVHD associated with Tacrolimus and Mycophenolate Mofetil as post-grafting immunosuppression.

OTHER OUTCOMES:
Survival | Post 100 days
  Overall survival will be followed

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Brunvand, MD, Principal Investigator — Colorado Blood Cancer Institute
Locations (1):
- Colorado Blood Cancer Institute, Denver, Colorado, United States